CLINICAL TRIAL: NCT01661933
Title: Combining Necator Americanus With Trace Gluten to Restore Tolerance in Coeliac Disease: a Pilot Clinical and a Detailed in Vitro Immunological Study.
Brief Title: Desensitising Celiac Disease Patients With the Human Hookworm
Acronym: NaCeD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Prince Charles Hospital (Other Government)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Principal Investigator, Dr John Croese, Chief Investigator, The Prince Charles Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: AU/3/BOBD012
Record Dates: First submitted 2012-08-06; First posted 2012-08-10 (Estimated); Results first posted 2014-10-13 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Celiac Disease
Keywords: celiac disease; hookworm; probiotic
MeSH Terms: conditions — Celiac Disease; Ancylostomiasis | interventions — ASP-1 protein, Necator americanus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Necator americanus, gluten challenge (Experimental): Single arm, vertical.
  Interventions: Biological: Necator americanus

INTERVENTIONS:
Biological: Necator americanus — Previously inoculated subjects will be further inoculated as previously undertaken with 20 3rd stage infective Na larvae (10 + 10 over 4 weeks). Four weeks after the 2nd inoculation, each participant will receive a micro-dose of gluten (10 mg daily) as pasta for 8 weeks, to be followed by a low-dose of gluten (50 mg daily) for 8 weeks. After this, a detailed assessment involving upper endoscopy and duodenal biopsy will be performed before deciding on an individual case basis that it is safe for the participant to proceed to challenge. A gluten challenge of 1 G (15-20 G of pasta or a ½ slice of standard white bread) twice weekly for 12 weeks will commence.
  Other Names: Hookworm
Biological: Necator americanus — After completion of the previously planned challenge, volunteers will be invited to extend the gluten challenge. The extension is for 4 weeks total. The gluten challenge is stepwise: gluten 10 mg daily for one week, 50 mg daily for one week and finally 3 grams daily for 2 weeks. The outcome measure is serum tissue transglutaminase to be compared before and after the intervention.
  Other Names: Hookworm

SUMMARY:
We have established that the hookworm Necator americanus (Na) dramatically alters the local and systemic immune landscape of the infected human host. Consistent with the principle of desensitisation, diet managed celiac disease subjects previously infected by us with Na will be invited to receive small incremental doses of gluten as pasta (3-25 mm straw of spaghetti) over 16 weeks. Each participant will then be carefully re-assessed to determine if it is appropriate to undertake a 12-week gluten challenge.

DETAILED DESCRIPTION:
Hypothesis The adaptive Th2/regulatory profile imposed by Na will promote gluten tolerance following a micro-dose desensitising programme.

Primary Aim: To determine the safety and efficacy of Na as a tolerising agent in celiac subjects

Specific Aim 1. Undertake a therapeutic pilot study comparing mucosal histopathology before and after a gluten challenge, to be preceded by a programmed desensitising micro-challenge using Na as a tolerising agent.

Specific Aim 2. Assess systemic and mucosal immune responses to gluten micro-challenge, Na infection, and gluten re-challenge throughout the pilot study, to be referenced against hookworm-naive people with treated and untreated celiac disease.

Specific Aim 3. Utilising blood and tissue from hookworm-naive celiac disease volunteers, undertake in vitro studies focusing on the effects of Na-derived excretory/secretory (ES) products on gluten-stimulated gut mucosal cell apoptosis, cytokine and gene profiles.

ELIGIBILITY:
Inclusion Criteria:

* Previously enrolled adults who received an experimental hookworm infection with diet treated celiac disease.

Exclusion Criteria:

* Immune suppressive therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-08; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Croese, MD, Study Director — The Prince Charles Hospital, Centre for Biodiscovery and Molecular Development of Therapeutics; Dianne Jones, BAppSc, Principal Investigator — Logan Hospital; Alexander Loukas, PhD, Principal Investigator — Centre for Biodiscovery and Molecular Development of Therapeutics, James Cook University
Locations (1):
- Prince Charles Hospital, Chermside, Queensland, Australia

REFERENCES:
- [Background] Daveson AJ, Jones DM, Gaze S, McSorley H, Clouston A, Pascoe A, Cooke S, Speare R, Macdonald GA, Anderson R, McCarthy JS, Loukas A, Croese J. Effect of hookworm infection on wheat challenge in celiac disease--a randomised double-blinded placebo controlled trial. PLoS One. 2011 Mar 8;6(3):e17366. doi: 10.1371/journal.pone.0017366. PMID 21408161

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 20 potential candidates, 2 could not be contacted (address changed), 1 was not interested, and 5 were unavailable (travel-2, pregnancy-2 or study-1 commitments). Twelve enrolled in September 2012. 8 committed to 3 endoscopic procedures and 2 committed to two endoscopies.
Groups:
- Necator Americanus, Gluten Challenge: Single arm, vertical. Necator americanus: Subjects were inoculated with 20 3rd stage Na larvae (10 + 10 over 4-8 weeks). After hookworm colonization, a micro-dose gluten challenge of 10 mg daily for 6 weeks, followed by 50 mg daily for 6 weeks was completed. After this, a detailed assessment including histology was performed to establish it safe for the participant to proceed to a low-dose gluten challenge of 25 mg daily and 1 G (15-20 G of pasta) twice weekly for 12 weeks. After low-dose challenge, a further evaluation was undertaken before inviting participants to undertake a gluten challenge of 3 G daily over for 2 weeks (preceded by a micro-dose 2 week lead-in).
Period: Gluten Micro-challenge
Arm/Group | Necator Americanus, Gluten Challenge
Started | 12 (All 12 enrolled completed hookworm inoculation and gluten micro-challenge.)
Completed | 12 (Two gluten intolerant participants did not proceed to the low-dose challenge.)
Not Completed | 0
Period: Low-dose Gluten Challenge
Arm/Group | Necator Americanus, Gluten Challenge
Started | 12 (One was symptomatically intolerant to gluten >25 mg. One had active CeD pre- & post-micro-challenge)
Completed | 10 (Two had challenge interrupted for 1-2 weeks. All completed challenge.)
Not Completed | 2
Not completed — Physician Decision | 2
Period: High-dose Gluten Challenge
Arm/Group | Necator Americanus, Gluten Challenge
Started | 10 (2 of 10 available after post-GC-1g did not enroll for reasons unrelated to gluten.)
Completed | 8
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Mean age 53 years, range 39-67; females 9.
Groups:
- Gluten Micro-challenge: Single arm, vertical. All twelve healthy adults enrolled subjects were successfully inoculated with hookworm and there was no serious adverse response. Individual hemoglobin levels were all normal and the group mean had significantly increased unexpectedly at completion of the study. Histology was not graded until after low-dose challenge but retrospectively confirmed enrollment Marsh scores of M0-8, M1-1, M2-2 and M3a-1. All participants were complying with a gluten-free diet, were symptomatically well and had a normal anti-tTG.
Arm/Group | Gluten Micro-challenge
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 53 [39 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Duodenal Villus Height:Crypt Depth
Description: Biopsies were fixed in neutral buffered formalin, processed and carefully orientated and embedded in paraffin wax. Sections (3 µm) were stained with H&E. Slides from both time-points were de-identified, shuffled and graded by Dr John Croese after which results from poorly orientated slides were verified by Dr Andrew Clouston. The Vh:Cd ratios were measured on 5 randomly selected well-orientated sites. The null hypothesis is that hookworm infection will not protect against mucosal damage following 12-week exposure to gluten in celiac disease.
Time Frame: Week -24 to -36
Population: All 10 of 12 participants who completed micro-challenge successfully progressed and completed low-dose challenge.
Measure: Mean (95% Confidence Interval); unit: Ratio
Groups:
- Necator Americanus, Gluten Challenge: Single arm, vertical. Necator americanus: Subjects were inoculated with 20 3rd stage Na larvae (10 + 10 over 4-8 weeks). After hookworm colonization, a micro-dose gluten challenge of 10 mg daily for 6 weeks, followed by 50 mg daily for 6 weeks was completed. After this, assessments including histology were performed to establish it safe for the participant to proceed to a low-dose gluten challenge of 25 mg daily and 1 G (15-20 G of pasta) twice weekly for 12 weeks. After low-dose challenge, a further evaluation was undertaken before inviting participants to undertake a gluten challenge of 3 G daily over for 2 weeks (preceded by a micro-dose 2 week lead-in).
Arm/Group | Necator Americanus, Gluten Challenge
Number analyzed (Participants) | 10
Ratio
  Baseline | 2.73 [2.31 to 3.15]
  Low-dose gluten | 2.73 [2.31 to 3.15]
Statistical Analysis 1: Comparison: Necator Americanus, Gluten Challenge; Test type: Superiority or Other; p = 0.693, t-test, 2 sided

2. Secondary Outcome: Intraepithelial Lymphocyte Count
Description: Biopsies were fixed in neutral buffered formalin, processed and carefully orientated and embedded in paraffin wax. Sections (3 µm) were stained with anti-CD3. All slides were de-identified and graded by Dr John Croese. The IEL percentages were measured on 2 or more randomly selected well-orientated villi. The null hypothesis is that hookworm infection will not protect against mucosal IEL influx following 12-week exposure to gluten in celiac disease.
Time Frame: Week-24 and -36
Measure: Mean (95% Confidence Interval); unit: Percentage of epithelial cells
Arm/Group | Necator Americanus, Gluten Challenge
Number analyzed (Participants) | 10
Percentage of epithelial cells
  Baseline | 33.40 [27.12 to 39.68]
  Low-dose gluten | 35.00 [28.72 to 41.28]
Statistical Analysis 1: Comparison: Necator Americanus, Gluten Challenge; Test type: Superiority or Other; p = 0.837, t-test, 2 sided

3. Secondary Outcome: Number of Participants With 2 Points Increase in Marsh Score Post GC-1g
Description: The Marsh score is a defined but qualitative assessment assigned a value to allow for comparison. The scores were evaluated by consensus between the primary (chief) investigator and the study pathologist. The Marsh score was graded 0, 1, 2, 3A (assigned-4), 3B (-5) and 3C (-6); rage 1-6 with normal=0 and severe inflammation=6. Because the scoring is vulnerable to artefact, only a 2-point shift was regarded as a significant intra-individual change. The scores were graded after week-36 on biopsies de-identified shuffled. An upward shift was interpreted to reflect a significant worsening of gluten-associated inflammation. The comparison reported evaluated changes from baseline (week-24) to post-low-dose gluten challenge (week-24; GC-1g). The objective for using the Marsh score was to identify individuals who might have experienced a severe worsening in pathology due to GC-1g that might not be reflected in the Vh:Cd group analysis.
Time Frame: Longitudinal change between week-24 and week-36
Population: The outcome score was the number with a 2-point increase in Marsh 3 score post GC-1g.
Measure: Number; unit: participants
Groups:
- Necator Americanus, Pre-gluten Challenge: Single arm, vertical. Ten of 12 participants enrolled based on symptomatic tolerance of gluten and satisfactory histology during and after micro-challenge. 2 were withdrawn pre-GC-1g, one who was symptomatically intolerant of gluten and one who had M3a after micro-challenge. Pre-GC1g scores.
Arm/Group | Necator Americanus, Pre-gluten Challenge
Number analyzed (Participants) | 10
participants | 1
Statistical Analysis 1: Comparison: Necator Americanus, Pre-gluten Challenge; The null hypothesis was that irrespective of hookworm infection, GC-1g would result in a 2-point or more deterioration in the Marsh score. A binomial (yes=deterioration or no=no deterioration) distribution was applied to pre- and post-GC-1g paired biopsies; Test type: Superiority or Other; p = 0.99, Binomial distribution

4. Secondary Outcome: Serum Anti-tissue Transglutaminase Antibodies Measured as International Units/mL (IU/mL)
Description: The trial was extended with pre-trial and mid-trial anti-tTG antibody levels used to compare with the post-trial levels. Anti-tTG is a serological measure of tissue transglutaminase-2 antibodies. In active celiac disease, levels are increased. In treated disease, levels are low (normal cut-off was <15 IU/mL). A significant increase compared to baseline in tTG can be expected 2 weeks after consuming 3g of gluten daily for 2 weeks in people with celiac disease who have been maintaining a gluten-free diet, but who are not taking other treatment.
Time Frame: Anti-tTG IU/mL levels pre-trial, mid-trial and after 3 gram/day gluten challenge
Population: 2 of 12 participants did not progress past baseline micro-challenge, 2 of 10 participants did not progress past low-dose challenge.
Measure: Mean (95% Confidence Interval); unit: International Units/mL
Arm/Group | Necator Americanus, Gluten Challenge
Number analyzed (Participants) | 8
International Units/mL
  Baseline | 4.12 [3.12 to 5.10]
  Low-dose gluten | 2.99 [2.00 to 3.94]
  After 3 G gluten daily | 2.11 [1.16 to 3.07]
Statistical Analysis 1: Comparison: Necator Americanus, Gluten Challenge; Test type: Superiority or Other; p = 0.005, Mixed effects model

ADVERSE EVENTS:
Groups:
- Gluten Micro-challenge: Single arm, longitudinal study of responses to escalating gluten doses in people with celiac disease after infection with Necator americanus, a human hookworm.
Arm/Group | Gluten Micro-challenge
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 2/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gluten Micro-challenge (N=12)
Symptomatic gluten intolerance (Gastrointestinal disorders) | 1 (1) — One subject experienced nausea and pain when gluten doses exceeded 25 mg/d and was advised not to continue.
Active CeD (Gastrointestinal disorders) | 1 (1) — One subject had Marsh 3a inflammation on biopsy collected immediately post-micro-challenge. Retrospective analysis established that this was likely present immediately pre-trial.

LIMITATIONS AND CAVEATS:
Open study. Small number. Historical controls.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No